CLINICAL TRIAL: NCT03369756
Title: A Prospective Study of Quality of Life in Patients With Chronic Leg Wound(s) Treated With Prontosan® Wound Irrigation Solution and Prontosan® Wound Gel
Brief Title: Prontosan Quality of Life Study in Patients With Chronic Leg Wound(s)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated due to prolonged subject recruitment
Sponsor: B. Braun Medical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OPM-G-H-1506
Record Dates: First submitted 2017-12-06; First posted 2017-12-12 (Actual); Results first posted 2020-12-08 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-11

CONDITIONS: Wound of Lower Leg (Physical Finding)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Prontosan Solution and Gel (Other): Treatment with Prontosan® Wound Irrigation Solution and Prontosan® Wound Gel over 4 week period
  Interventions: Device: Prontosan Wound Irrigation Solution and Prontosan Wound Gel

INTERVENTIONS:
Device: Prontosan Wound Irrigation Solution and Prontosan Wound Gel — Wound cleansing using Prontosan solution and gel

SUMMARY:
This study evaluates the use of Prontosan® Wound Irrigation Solution and Prontosan® Wound Gel in the treatment of chronic leg wounds in adults. All participants will use Prontosan and report their personal observations regarding Quality of Life.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥18 years of age
2. Either 2 wounds on 1 leg or 1 wound on each leg or only 1 wound. Wound(s) must be located below the knee.
3. At least one wound must have a surface area ≥5 cm2 and ≤50 cm2 and it also must be present for ≥4 weeks
4. Mean global score ≥1.18 on the Wound-QoL questionnaire (this will be calculated by the electronic data capture [EDC] system at the time of screening to assess eligibility)
5. Willingness to wear an off-loading device if medically indicated (e.g., DH shoe or walker)

Exclusion Criteria:

1. Prior treatment with Prontosan solution or Prontosan gel on the wound(s)
2. Infection in the wound(s)
3. Cartilage exposure in the wound(s)
4. Antibiotic therapy within 7 days prior to baseline (i.e., prior to first administration of study treatment). Topical antibiotics not applied to the wound are acceptable.
5. Current diagnosis of severe peripheral artery disease as indicated by clinical findings (i.e., no palpable pulse on both dorsal pedis and posterior tibial arteries of the affected limb) or an Ankle Brachial Index of < 0.5
6. Presence of gangrene in the wound(s) or on the leg(s)
7. Active (flare up) rheumatic or collagen vascular disease (including rheumatoid arthritis, scleroderma, and systemic lupus erythematosus), psoriasis, sarcoidosis, or other skin disease. These subjects are allowed to receive oral, inhaled, or parenteral corticosteroids, immunosuppressive agents, or cytotoxic agents. Note: fibromyalgia is acceptable.
8. Osteomyelitis diagnosed by x-ray, bone biopsy, or other radiological procedure within 90 days prior to the screening visit
9. Active radiation therapy below the hip
10. Subjects with medical conditions other then those identified in Exclusion Criteria 7 who are currently receiving or has received oral, or parenteral corticosteroids, immunosuppressive agents, or cytotoxic agents within 30 days prior to baseline (i.e., prior to first administration of study treatment) or is anticipated to require such agents during the course of the study
11. Clinical laboratory values that may impair wound healing; for example, hemoglobin <10 g/dL, or HbA1c ≥12%
12. Enrolled in any investigational drug or device study for any disease/indication within 30 days prior to the screening visit
13. Unable to comprehend or comply with study requirements, or inability to sign an informed consent form
14. Allergic to any of the components in Prontosan solution or Prontosan gel
15. Patients who, in the opinion of the Investigator, would not be suitable candidates for this study or have some impediment to their ability to heal
16. Preplanned surgery or procedures that would occur during the study (other than deemed minor and clinically non-significant by the Investigator) or that would interfere with the study
17. Phase 4 pressure ulcer as defined by full-thickness skin and tissue loss with exposed or directly palpable fascia, muscle, tendon, ligament, cartilage or bone in the ulcer. Slough and/or eschar may be visible
18. Severe secondary lymphedema as diagnosed by clinical findings in inferior members (e.g., legs)
19. A diagnosis of malnutrition as determined by either a low BMI (<18.5 kg/m2), or on the combined finding of weight loss together with reduced BMI (age-specific)
20. Employee of the Investigator or study center, with direct involvement in the study or other studies under the direction of that Investigator or study center, as well as family members of the employees or the Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2019-09-25 (Actual); Study Completion 2019-09-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Jupiter Medical Center, Jupiter, Florida
  - Barry University Clinical Research, North Miami Beach, Florida
  - Northwell Comprehensive Wound Care Healing Center and Hyperbarics, North New Hyde Park, New York
  - St. Luke's Wound Care Center, Bethlehem, Pennsylvania
  - Harrisburg Foot and Ankle Center, Harrisburg, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Richmond NA, Maderal AD, Vivas AC. Evidence-based management of common chronic lower extremity ulcers. Dermatol Ther. 2013 May-Jun;26(3):187-96. doi: 10.1111/dth.12051. PMID 23742279
- [Background] Frykberg RG, Banks J. Challenges in the Treatment of Chronic Wounds. Adv Wound Care (New Rochelle). 2015 Sep 1;4(9):560-582. doi: 10.1089/wound.2015.0635. PMID 26339534
- [Background] McCarty SM, Percival SL. Proteases and Delayed Wound Healing. Adv Wound Care (New Rochelle). 2013 Oct;2(8):438-447. doi: 10.1089/wound.2012.0370. PMID 24688830
- [Background] Leaper DJ, Schultz G, Carville K, Fletcher J, Swanson T, Drake R. Extending the TIME concept: what have we learned in the past 10 years?(*). Int Wound J. 2012 Dec;9 Suppl 2(Suppl 2):1-19. doi: 10.1111/j.1742-481X.2012.01097.x. PMID 23145905
- [Background] Romanelli M, Dini V, Barbanera S, Bertone MS. Evaluation of the efficacy and tolerability of a solution containing propyl betaine and polihexanide for wound irrigation. Skin Pharmacol Physiol. 2010;23 Suppl:41-4. doi: 10.1159/000318266. Epub 2010 Sep 8. PMID 20829661
- [Background] Andriessen AE, Eberlein T. Assessment of a wound cleansing solution in the treatment of problem wounds. Wounds. 2008 Jun;20(6):171-5. PMID 25942522
- [Background] Blome C, Baade K, Debus ES, Price P, Augustin M. The "Wound-QoL": a short questionnaire measuring quality of life in patients with chronic wounds based on three established disease-specific instruments. Wound Repair Regen. 2014 Jul-Aug;22(4):504-14. doi: 10.1111/wrr.12193. PMID 24899053
- [Background] Augustin M, Baade K, Herberger K, et al. Use of the Wound-QoL instrument in routine practice: feasibility, validity, and development of an implementation tool. Wound Medicine. 2014;5:4-8
- See also: Wound-QoL Short Manual, dated September 2015 — http://www.wound-qol.com
- See also: Measuring wounds on Wound Care Advisor — http://woundcareadvisor.com/measuring-wounds

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Prontosan Solution and Gel
Started | 43
Completed | 36 (36 completed 4 weeks of treatment; 40 were considered statistical completers)
Not Completed | 7

BASELINE CHARACTERISTICS:
Arm/Group | Prontosan Solution and Gel
Number analyzed (Participants) | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.2 (15.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 15
  White | 17
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 36

OUTCOME MEASURES:

1. Primary Outcome: Wound-QoL Global Score
Description: The Wound-QoL is a tool to measure disease-specific, health-related quality of life of patients with chronic wounds. It consists of 17 items on impairments which is assessed for the previous 7 days and is competed by the patient. It has 3 subscales that can assess "Body", "Psyche" and "Everyday Life". These subscales cover items 1 to 16. Item 17 is not part of any of the subscales. The Wound-QoL can be used in clinical and observational studies and in daily practice.
  Each individual item is rated on a scale ranging from 0 (not at all) to 4 (very much). A "Total" or "Global" score is the average of at least 13 completed questions, regardless of which questions were not completed. The average of each of the 3 subscales can be computed if no more than 1 item of the subscale is missing. The higher values represents more of an impact to the patient for that item.
Time Frame: 5 weeks overall (4 weeks of treatment and/or observations followed by a one-day visit at end of study in week 5)
Population: All subjects who completed 4 weeks of treatment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prontosan Solution and Gel
Number analyzed (Participants) | 36
score on a scale
  Week 1 / Baseline | 2.41 (0.99)
  Week 2 | 1.74 (1.15)
  Week 3 | 1.51 (0.95)
  Week 4 | 1.25 (0.90)
  Week 5 / End | 1.30 (0.87)

2. Secondary Outcome: Wound QoL Subscore; Body Dimension
Description: The Wound-QoL is a tool to measure disease-specific, health-related quality of life of patients with chronic wounds. It consists of 17 items on impairments which is assessed for the previous 7 days and is competed by the patient. It has 3 subscales that can assess "Body", "Psyche" and "Everyday Life". It can be used in clinical and observational studies and in daily practice.
  Subscale "Body" consists of Items #1 to #5. Each individual item is rated on a scale ranging from 0 (not at all) to 4 (very much). The average of the subscale can be computed if no more than 1 item of the subscale is missing. The higher values represents more of an impact to the patient for that item.
Time Frame: 5 weeks overall (4 weeks of treatment and/or observations followed by a one-day visit at end of study in week 5)
Population: All subjects who completed 4 weeks of treatment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prontosan Solution and Gel
Number analyzed (Participants) | 36
score on a scale
  Body Subscore change, Baseline / Week 1 to Week 2 | -0.76 (1.15)
  Body Subscore change, Baseline / Week 1 to Week 3 | -0.93 (1.28)
  Body Subscore change, Baseline / Week 1 to Week 4 | -1.19 (1.30)
  Body Subscore change, Baseline / Week 1 to End / Week 5 | -1.17 (1.21)

3. Secondary Outcome: Wound QoL Subscore; Psyche Dimension
Description: The Wound-QoL is a tool to measure disease-specific, health-related quality of life of patients with chronic wounds. It consists of 17 items on impairments which is assessed for the previous 7 days and is competed by the patient. It has 3 subscales that can assess "Body", "Psyche" and "Everyday Life". It can be used in clinical and observational studies and in daily practice.
  Subscale "Psyche" consists of Items #Items #6 to #10. Each individual item is rated on a scale ranging from 0 (not at all) to 4 (very much). The average of the subscale can be computed if no more than 1 item of the subscale is missing. The higher values represents more of an impact to the patient for that item.
Time Frame: 5 weeks overall (4 weeks of treatment and/or observations followed by a one-day visit at end of study in week 5)
Population: All subjects who completed 4 weeks of treatment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prontosan Solution and Gel
Number analyzed (Participants) | 36
score on a scale
  Psyche Subscore change, Baseline / Week 1 to Week 2 | -0.77 (1.12)
  Psyche Subscore change, Baseline / Week 1 to Week 3 | -1.04 (1.13)
  Psyche Subscore change, Baseline / Week 1 to Week 4 | -1.24 (1.27)
  Psyche Subscore change, Baseline / Week 1 to End / Week 5 | -1.26 (1.14)

4. Secondary Outcome: Wound QoL Subscore; Everyday Life Dimension
Description: The Wound-QoL is a tool to measure disease-specific, health-related quality of life of patients with chronic wounds. It consists of 17 items on impairments which is assessed for the previous 7 days and is competed by the patient. It has 3 subscales that can assess "Body", "Psyche" and "Everyday Life". It can be used in clinical and observational studies and in daily practice.
  Subscale "Everyday Life" consists of Items #Items #11 to #16. Each individual item is rated on a scale ranging from 0 (not at all) to 4 (very much). The average of the subscale can be computed if no more than 1 item of the subscale is missing. Generally, the higher values represents more of an impact to the patient for that item.
Time Frame: 5 weeks overall (4 weeks of treatment and/or observations followed by a one-day visit at end of study in week 5)
Population: All subjects completing 4 weeks of treatment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prontosan Solution and Gel
Number analyzed (Participants) | 36
score on a scale
  Everyday Life Subscore change, Baseline / Week 1 to Week 2 | -0.58 (1.05)
  Everyday Life Subscore change, Baseline / Week 1 to Week 3 | -0.82 (1.04)
  Everyday Life Subscore change, Baseline / Week 1 to Week 4 | -1.11 (1.11)
  Everyday Life Subscore change, Baseline / Week 1 to End / Week 5 | -1.00 (0.99)

5. Other Pre Specified Outcome: Wound Size
Description: Change in wound size from Baseline/Week 1 to Final/Week 5. The change in the size of a wound will be evaluated using a disposable ruler to directly measure the overall wound dimensions at each scheduled visit to the study site (Weeks 1 and 5). These measurements will be done before any cleaning of the wound and after cleaning the wound (debridement).
Time Frame: 5 weeks overall (4 weeks of treatment and/or observations followed by a one-day visit at end of study in week 5)
Population: All subjects who completed 4 weeks of treatment.
Measure: Mean (Standard Deviation); unit: wound surface area (cm^2)
Arm/Group | Prontosan Solution and Gel
Number analyzed (Participants) | 36
wound surface area (cm^2)
  Pre-Debridement Wound Size Change (Baseline/Week 1 to Week 5 / End): number analyzed (Participants) | 35
  Pre-Debridement Wound Size Change (Baseline/Week 1 to Week 5 / End) | -6.6 (18.3)
  Post-Debridement Wound Size Change(Baseline/Week 1 to Final/Week 5): number analyzed (Participants) | 31
  Post-Debridement Wound Size Change(Baseline/Week 1 to Final/Week 5) | -8.2 (19.2)

ADVERSE EVENTS:
Time Frame: Screening through 4th week of treatment (5 weeks total).
Description: All reported adverse events were recorded. It was decided that only Prontosan related AEs, all SAEs, and ADEs would be coded by the Sponsor according to the final version of the SAP (v2.0 dated 04-Nov-2019).
Arm/Group | Prontosan Solution and Gel
All-Cause Mortality (participants affected / at risk) | 0/43
Serious Adverse Events (participants affected / at risk) | 5/43
Other Adverse Events (participants affected / at risk) | 14/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prontosan Solution and Gel (N=43)
Back Pain (General disorders) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Compression Fracture (Injury, poisoning and procedural complications) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prontosan Solution and Gel (N=43)
Burning Sensation (General disorders) | 11 (62)
Pain (General disorders) | 3 (13)
Paraesthesia (General disorders) | 1 (1)
Burning Sensation (Skin and subcutaneous tissue disorders) | 1 (1)
Pain (Skin and subcutaneous tissue disorders) | 1 (1)
Pain of Skin (Skin and subcutaneous tissue disorders) | 1 (10)
Paraesthesia (Skin and subcutaneous tissue disorders) | 4 (18)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (4)
Sensitive Skin (Skin and subcutaneous tissue disorders) | 1 (1)
Skin Disorder (Skin and subcutaneous tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
All reported adverse events were recorded. It was decided that only Prontosan related AEs, all SAEs, and ADEs would be coded by the Sponsor according to the final version of the SAP (v2.0 dated 04-Nov-2019).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution acknowledges and shall cause Investigator to acknowledge that Sponsor has the right to use the Study Results in any manner deemed appropriate to Sponsor's business interests, both during, and following termination of, this Agreement. Where Institution and/or Investigator require the use of the Study Results for publication, the Institution and/or Investigator shall seek the Sponsor's written approval which shall not be unreasonably withheld.

DOCUMENTS (3):
  • Study Protocol (2018-11-14): https://cdn.clinicaltrials.gov/large-docs/56/NCT03369756/Prot_000.pdf
  • Informed Consent Form (2017-09-21): https://cdn.clinicaltrials.gov/large-docs/56/NCT03369756/ICF_001.pdf
  • Statistical Analysis Plan (2019-11-04): https://cdn.clinicaltrials.gov/large-docs/56/NCT03369756/SAP_002.pdf